CLINICAL TRIAL: NCT00880217
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group, Multicenter Study of 3 Dosages of JNJ-31001074 in the Treatment of Adult Subjects With Attention-Deficit/Hyperactivity Disorder
Brief Title: A Study to Evaluate 3 Different Doses of JNJ-31001074 in the Treatment of Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015964; 31001074ATT2001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders with Hyperactivity; Adult ADHD; JNJ-31001074
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; bavisant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 001 (Experimental): JNJ-31001074 1 mg/d 1-mg capsule once daily for 42 days
  Interventions: Drug: JNJ-31001074 1 mg/d
- 002 (Experimental): JNJ-31001074 3 mg/d 3-mg capsule once daily for 42 days
  Interventions: Drug: JNJ-31001074 3 mg/d
- 003 (Experimental): JNJ-31001074 10 mg/d 10-mg capsule once daily for 42 days
  Interventions: Drug: JNJ-31001074 10 mg/d
- 004 (Active Comparator): Atomoxetine 80 mg/d 40-mg capsule for 3 days followed by 80-mg capsule once daily for 39 days
  Interventions: Drug: Atomoxetine 80 mg/d
- 005 (Active Comparator): OROS methylphenidate HCl 54 mg/d 36-mg capsule for 3 days followed by 54-mg capsule once daily for 39 days
  Interventions: Drug: OROS methylphenidate HCl 54 mg/d
- 006 (Placebo Comparator): Placebo capsule once daily for 42 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine 80 mg/d — 40-mg capsule for 3 days, followed by 80-mg capsule once daily for 39 days
  Arms: 004
Drug: Placebo — Placebo capsule once daily for 42 days
  Arms: 006
Drug: OROS methylphenidate HCl 54 mg/d — 36-mg capsule for 3 days, followed by 54-mg capsule once daily for 39 days
  Arms: 005
Drug: JNJ-31001074 3 mg/d — 3-mg capsule once daily for 42 days
  Arms: 002
Drug: JNJ-31001074 1 mg/d — 1-mg capsule once daily for 42 days
  Arms: 001
Drug: JNJ-31001074 10 mg/d — 10-mg capsule once daily for 42 days
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety/tolerability of 3 different dosages of JNJ-31001074 compared with placebo in adult patients with attention-deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
This will be a randomized (study drug assigned by chance), double-blind (neither the investigator nor the patient know the name of the assigned study drug), placebo- and active-controlled, parallel-group, multicenter study in patients with adult ADHD. The study population will include approximately 426 male and female patients, 18 to 55 years of age (inclusive) with a DSM-IV diagnosis of ADHD, who will be randomly assigned (like flipping a coin) in a 1:1:1:1:1:1 ratio to 1 of 6 treatment groups (1 milligrams per day [mg/d] JNJ-31001074, 3 mg/d JNJ-31001074, 10 mg/d JNJ 31001074, 80 mg/d atomoxetine HCl, 54 mg/d controlled-release [OROS] methylphenidate HCl, or placebo). Study centers will make every attempt to include approximately 4 women for every 10 men randomized. The study will consist of 3 phases: a screening phase of up to 7 days; a 42-day double-blind treatment phase; and a 7-day post-treatment phase, in which the investigator staff will call patients 7 days after the last dose of study drug, to ask about any adverse events. The total duration of patient participation will be approximately 8 weeks. During the screening and double-blind treatment phases, patients will have periodic assessments at visits (screening, Day 1, Day 4, Day 7, Day 14, Day 28, and Day 42) of the following: severity of ADHD symptoms, including inattention and impulsivity; daily function; sleep experience; and cigarette consumption and cigarette craving. In addition, patients will be asked to include an adult household member to complete the observer version of the Conners Adult ADHD Rating Scale (CAARS-O:SV) at the beginning and end of the study. Patients will take one oral capsules each day in the morning upon awakening, either JNJ-31001074 (1, 3, or 10 mg), matching atomoxetine HCL (40 or 80 mg), matching OROS methylphenidate HCl (36 or 54 mg), or matching placebo. For atomoxetine HCl, patients will receive 40 mg/d for the first 3 days, and 80 mg/d for the remainder of the study. For OROS methylphenidate HCl, patients will receive 36 mg/d for the first 3 days, and 54 mg/d for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ADHD, confirmed with the Conners Adult ADHD Diagnostic Interview for Diagnostic and Statistical Manual, 4th edition (DSM-IV) (CAADID)
* Patients who meet the cutoff scores for the Conners Adult ADHD Rating Scale (CAARS-S:SV)
* Patients with a Clinical Global Impression - Severity (CGI-S) score of >=4 out of 7
* Patients must have a body mass index between 18.0 and 35.0 (inclusive)
* Women must be postmenopausal for >=2 years, surgically sterile, abstinent, or practice a double-barrier method of birth control in addition to any other forms of birth control
* Women of childbearing potential must have a negative pregnancy test at screening
* Men must agree to use a double-barrier method of birth control and to not donate sperm during the study and for 3 months after the last dose of study drug
* Female partners of male patients must be postmenopausal, surgically sterile, abstinent, or also use an effective method of birth control.

Exclusion Criteria:

* Patients with any current Axis I psychiatric disorder
* Patients with a diagnosis of autism or Asperger's syndrome
* Patients with motor tics or a family history or diagnosis of Tourette's syndrome
* Patients with a diagnosis of a primary sleep disorder
* Patients who are suicidal or have previously attempted suicide
* Patients with a history of substance abuse or dependence within 6 months prior to screening
* Patients who have taken any mood stabilizer, antipsychotic, antidepressant, or anxiolytic within 3 months prior to screening
* Patients who have started behavioral or cognitive behavioral therapy specifically for ADHD within 3 months prior to screening
* Patients who have not responded previously to treatment with a psychostimulant medication or to treatment with atomoxetine HCl or OROS methylphenidate HCl.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 430 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the ADHD rating scale total score | Through Day 42

SECONDARY OUTCOMES:
Secondary endpoints will include Clinical Global Impression of Change (CGI-C). | At the end of the double-blind treatment phase (Day 42)
Other secondary endpoints will include the change from baseline in the Conners Adult ADHD Rating Scale (CAARS-S:SV) and the Clinical Global Impression - Severity (CGI-S). | Through the end of the double-blind treatment phase (Day 42)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (35):
- United States (35):
  - Little Rock, Arkansas
  - Lafayette, California
  - Los Alamitos, California
  - Santa Ana, California
  - Wildomar, California
  - Bradenton, Florida
  - Jacksonville, Florida
  - North Miami, Florida
  - Orlando, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Eagle, Idaho
  - Libertyville, Illinois
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Rochester Hills, Michigan
  - Saint Charles, Missouri
  - Mount Kisco, New York
  - New York, New York
  - Raleigh, North Carolina
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Media, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Wharton, Texas
  - Burlington, Vermont
  - Herndon, Virginia
  - Seattle, Washington
  - Middleton, Wisconsin

REFERENCES:
- [Derived] Weisler RH, Pandina GJ, Daly EJ, Cooper K, Gassmann-Mayer C; 31001074-ATT2001 Study Investigators. Randomized clinical study of a histamine H3 receptor antagonist for the treatment of adults with attention-deficit hyperactivity disorder. CNS Drugs. 2012 May 1;26(5):421-34. doi: 10.2165/11631990-000000000-00000. PMID 22519922